CLINICAL TRIAL: NCT00950105
Title: A Phase 1, Single Center, Randomized, Double-Blind, Placebo-Controlled Single Ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetic Profiles of Oral CPSI-2364 in Healthy Subjects
Brief Title: Single Ascending Dose Study of Oral CPSI-2364 (Semapimod)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 2364-CD-101
Record Dates: First submitted 2009-07-29; First posted 2009-07-31 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Crohn's Disease
Keywords: CPSI2364; Semapimod; Anti TNF alpha; Crohn's Disease; Safety; Tolerability; Pharmacokinetics
MeSH Terms: conditions — Crohn Disease | interventions — semapimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- CPSI-2364 1 mg p.o. (Experimental): Single dose
  Interventions: Drug: CPSI-2364 or placebo
- CPSI-2364 10 mg p.o. (Experimental): single dose
  Interventions: Drug: CPSI-2364 or placebo
- CPSI-2364 30 mg p.o. (Experimental): single dose
  Interventions: Drug: CPSI-2364 or placebo
- CPSI-2364 90 mg (Experimental): single dose
  Interventions: Drug: CPSI-2364 or placebo
- CPSI-2364 270 mg p.o. (Experimental): single dose
  Interventions: Drug: CPSI-2364 or placebo

INTERVENTIONS:
Drug: CPSI-2364 or placebo — Single, oral dose of CPSI-2364 or placebo
  Other Names: semapimod

SUMMARY:
This study will be conducted in healthy male or female subjects using a double-blind, randomized, placebo-controlled, single-dose design. Up to 30 subjects will be enrolled; 3 healthy subjects in Cohorts 1 and 2 (2 active, 1 placebo) and 8 healthy subjects in Cohorts 3 to 5 (6 active, 2 placebo). The following CPSI-2364 doses are proposed: 1 mg, 10 mg, 30 mg, 90 mg, and 270 mg.Safety will be evaluated throughout the study and include physical examinations, vital signs assessments, 12-lead electrocardiograms (ECGs), routine clinical laboratory tests (including blood chemistry, hematology, coagulation, and urinalysis), and adverse event (AE) assessments. Vital sign assessments and 12-lead ECGs will be performed repeatedly over the 24-hour observation period. Venous blood samples will be taken at specified intervals and tested for the presence of CPSI-2364.

DETAILED DESCRIPTION:
This study will be conducted in healthy male or female subjects using a double-blind, randomized, placebo-controlled, single-dose design. Up to 30 subjects will be enrolled; 3 healthy subjects in Cohorts 1 and 2 (2 active, 1 placebo) and 8 healthy subjects in Cohorts 3 to 5 (6 active, 2 placebo). The following CPSI-2364 doses are proposed: 1 mg, 10 mg, 30 mg, 90 mg, and 270 mg. In Cohort 1 (1 mg) and Cohort 2 (10 mg), the three subjects will all be dosed on the same day, with at least 60 minute intervals between dosing. In Cohorts 3 to 5, the first two subjects of each cohort (one active, one placebo) will receive their drug on the same day with at least a 60-minute interval between dosing, with the remainder of the cohort being dosed the next day once these subjects have been assessed. Safety labs, physical examination findings, and adverse events available up to and including Day 5 data of each cohort will be reviewed by the Investigator, the Study Manager, and the Sponsor (or designee) in order to determine the progression of dose escalation. Subjects will not be enrolled in the next higher cohort until the dose in the preceding cohort is deemed safe and tolerable. Doses will continue to be escalated in subsequent groups until a maximum tolerated dose (MTD) is reached, or until a top dose of 270 mg is reached, whichever is sooner. Intermediate and repeat dose levels may be administered in addition to or in place of the planned dose levels, if it is deemed appropriate to increase the safety or scientific value of this Phase 1 exploratory study.Safety will be evaluated throughout the study and include physical examinations, vital signs assessments, 12-lead electrocardiograms (ECGs), routine clinical laboratory tests (including blood chemistry, hematology, coagulation, and urinalysis), and adverse event (AE) assessments. Vital sign assessments and 12-lead ECGs will be performed repeatedly over the 24-hour observation period.Venous blood samples will be taken at specified intervals and tested for the presence of CPSI-2364.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria will be considered for admission to the study:

* male or female between 18 and 55 years old inclusive;
* for females, the following conditions are to be met: all female subjects must be confirmed as not pregnant via serum pregnancy test; females must be of non-childbearing potential (defined as either surgically sterile or at least 1 year postmenopausal); or female subjects of childbearing potential must use 2 of the 3 following acceptable birth control methods from the time specified prior to the study through 60 days following the last dose of study drug: intrauterine contraceptive device (IUD) in place for at least 2 months prior to study; barrier method (condom or diaphragm) with spermicide for at least 14 days prior to screening; stable hormonal contraceptive for at least 3 months prior to study;
* in good health as determined by the Investigator based on medical history, physical examination, ECG, and clinical laboratory tests;
* with a body mass index (BMI) of 19 to 30 kg/m2, inclusive;
* nonsmokers (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc., for 6 months prior to the administration of the study medication), subjects must have nicotine levels below those measured for smokers (less than 400 ng/mL);
* agrees to abstain from alcohol intake 48 hours before each administration of study agent and during inpatient portion of the study (Days -1 to 2);
* agrees to limit caffeine/methylxanthine (e.g., coffee, tea, chocolate, or caffeine-containing soft drinks) intake to less than 300 mg/day for the duration of the study (300 mg of caffeine is equal to approximately 3 cups of coffee or 6 cola drinks);
* agrees not to consume food or beverages containing grapefruit juice, Seville oranges, or quinine (e.g., tonic water) from 72 hours prior to study Day -1 until after the last PK sample is collected;
* capable of understanding and complying with the protocol; willing and able to adhere to the study visit schedule and other protocol requirements;
* have no relevant food allergies (e.g., eggs or other components of standard clinic meals); and
* must have signed the informed consent document prior to performance of any study related procedures.

Exclusion Criteria:

* currently have, or have a history of, disease or dysfunction of the renal, hepatic, pulmonary, cardiovascular, endocrine, hematologic, neurological, immune, gastrointestinal, genitourinary, or other body system, that is clinically significant in the opinion of the Investigator;
* likely hypersensitivity or allergies to CPSI-2364, any components of CPSI-2364, or any drug within the same class of drug, minor drug allergies to a drug in other drug class may be approved by the Investigator if not considered of clinical relevance;
* any subject with a clinically significant mental or physical illness (in the opinion of the Investigator/Medical Advisor) within 1 year prior to the first dose, including a history of alcohol and/or drug abuse (as defined by Diagnostic and Statistical Manual of Mental Disorders, 4th Edition guidelines) within 1 year prior to the first dose of study medication;
* abnormal pre-admission vital signs, 12-lead ECGs, and urinanalysis which are considered clinically significant by the Investigator and Sponsor (or designee);
* abnormal clinical laboratory evaluations, particularly abnormal creatinine, calculated GFR (abnormal defined as > 60 mL/min), and liver function tests. (Minor excursions from the normal range may be allowed if the clinical picture is otherwise normal and they are considered clinically insignificant by the Investigator and Sponsor [or designee]) ;
* any subject considering or scheduled to undergo any surgical procedure during the duration of the study;
* have an acute illness within 7 days prior to study agent administration or have had a hospitalization within 1 month prior to study agent administration;
* any subject who has received any known hepatic or renal clearance altering agents (eg, erythromycin, cimetidine, barbiturates, phenothiazines, or herbal/plant-derived preparations such as St. John's Wort, etc.) for a period of 90 days prior to the first dose of study medication;
* has a positive serology test for human immunodeficiency virus (HIV) antibodies, hepatitis A, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody at screening;
* has a positive urine drug screen for ethanol or substances of abuse including cocaine, cannabinoids, phencyclidine, amphetamines, benzodiazepines, barbiturates, opiates, propoxyphene, and methadone at screening and check-in(s);
* subject has donated plasma or blood within 30 days prior to the first dose of study medication or has a history of blood donation of more than 500 mL within 3 months prior to dosing;
* use of any prescription medications/products, except hormonal contraceptives, within 14 days prior to study entry, unless deemed acceptable by the Investigator;
* use of any over-the-counter (OTC) or nonprescription preparation (including minerals and phytotherapeutic/herbal/plant-derived preparations), within 14 days prior to dose administration, with the exception of ibuprofen and acetaminophen used at recommended doses. For acetaminophen a maximum of 1500 mg per day and no more than 3 g per week, will be allowed for the treatment of headache or other pain;
* any subject who does not meet the conditions for prior and concomitant treatments described in Section 8.8 Prior and Concomitant Therapy of this protocol;
* has taken any other investigational drug during the 30 days prior to Day -1;
* has any condition(s) that in the Investigator's opinion would: a) warrant exclusion from the study or b) prevent the subject from completing the study; or
* unable to understand verbal and/or written English or any other language in which a certified translation of the informed consent is available.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of CPSI-2364 | 7 days

SECONDARY OUTCOMES:
Pharmacokinetic profile of a single administration of oral CPSI-2364 | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Leese, MD, Principal Investigator — Quintiles Phase I unit, Overland Park, KS
Locations (1):
- Quintiles, Overland Park, Kansas, United States